CLINICAL TRIAL: NCT06399848
Title: Peritoneal Dialysis Daily Versus Six Days Per Week
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Timothy Meyer, Professor, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 75365
Record Dates: First submitted 2024-04-28; First posted 2024-05-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-05

CONDITIONS: Peritoneal Dialysis
MeSH Terms: interventions — SPHKAP protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peritoneal Dialysis Daily (Other): Each patient will compare their regular daily treatment with the effect of skipping a single day of treatment. There will be no other intervention.
  Interventions: Other: Skip one day of peritoneal dialysis treatment

INTERVENTIONS:
Other: Skip one day of peritoneal dialysis treatment — Skip one day of peritoneal dialysis treatment

SUMMARY:
The study will enroll patients receiving daily peritoneal dialysis who have significant residual native kidney function. The investiators will visit the patients at a routinely scheduled clinic visit and again at a non-routine visit after the patients skip a single day of dialysis. Blood samples will be obtained and a quality of life questionnaire will be administered at both visits.

The primary aim will be to determine whether the patients would prefer daily treatment or being allowed to skip one day per week.

Other aims will be to determine the effect of skipping a day on plasma levels of urea nitrogen and creatinine.

DETAILED DESCRIPTION:
The patients' preference will be assessed by asking the simple question would you prefer to perform peritoneal dialysis daily of six days per week.

The quality of life questionnaire to be used will be the Dialysis Symptom Index (DSI) which has a range of 0 to 150 with a high score reflecting worse quality of life.

The chemical to be measured will be the plasma urea nitrogen in mg/dl and the plasma creatinine in mg/dl as measured by the clinical laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Daily treament with peritoneal dialysis and residual native kidney funciton with residual urea clearance greater than 2 ml/min.

Exclusion Criteria:

* less than 3 months on peritoneal dialysis
* recent change in the dialysis prescriptoin
* recent peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Patient's preference for treatment regimen | Two weeks per patient
  Patient's stated preference for dialysis daily versus six days per week

SECONDARY OUTCOMES:
Symptoms | Two weeks per patient
  Quality of Life as assessed by a questionnaire
Plasma solute levels | Two weeks per patient
  Plasma levels of urea nitrogen and creatinine.

IPD SHARING:
Plan to Share IPD: No